CLINICAL TRIAL: NCT06818045
Title: Investigation of the Effect of Nonsurgical Periodontal Treatment Applied Together With Anti-TNF-α on Alveolar Bone Loss and Oxidative Stress in Patients With Rheumatoid Arthritis and Periodontitis
Brief Title: Nonsurgical Periodontal Treatment Combined With Anti-TNF-α in Patients With Rheumatoid Arthritis and Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hatice Yemenoğlu (Other)
Responsible Party: Sponsor-Investigator, Hatice Yemenoğlu, Principal investigator, Recep Tayyip Erdogan University Training and Research Hospital
Organization: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RecepTayyipErdogan University
Record Dates: First submitted 2025-02-02; First posted 2025-02-10 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-04

CONDITIONS: Peridontal Disease; Rheumatic Arthritis
Keywords: rheumatoid arthritis; periodontal disease; inflammation
MeSH Terms: conditions — Rheumatic Fever; Arthritis, Rheumatoid; Periodontal Diseases; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- control (Experimental)
  Interventions: Procedure: Non Surgical Periodontal Treatment; Other: Periodontal measurements will be performed; Other: biochemical measurements; Other: No medication will be administered to patients.

INTERVENTIONS:
Procedure: Non Surgical Periodontal Treatment — This procedure will be applied to all patients. All patients received nonsurgical periodontal treatment. Scaling root planing and subgingival debridement were performed.
Other: Periodontal measurements will be performed — Periodontal measurements will be performed on all patients (plaque index, gingival index, bleeding on probing, periodontal pocket depth, clinical attachment loss).
Other: biochemical measurements — Serum and gingival crevicular fluid (GCF) samples will be collected from patients for biochemical evaluations.
Other: No medication will be administered to patients. — No medication will be administered to patients.

SUMMARY:
Periodontitis is a multifactorial disease of the periodontium that can lead to destruction of the alveolar bone and supporting connective tissue and subsequent tooth loss. Recent studies have shown that periodontitis is associated with age, smoking habits, genetic predisposition, socioeconomic status, and various systemic diseases such as diabetes mellitus, atherosclerosis, obesity, osteoporosis, and rheumatoid arthritis (RA). RA is a chronic, systemic inflammatory disease of unknown etiology that primarily affects the joints. Periodontitis and RA have similar clinical and pathogenic features. Clinically, both diseases are characterized by local destruction of hard and soft tissues. Their pathogenesis involves the release of cytokines and matrix metalloproteinases (MMPs) from inflammatory cells. Expression of proinflammatory cytokines such as tumor necrosis factor-alpha (TNF-α) leads to the release of high levels of inflammatory mediators that cause bone destruction and the spread of inflammation. TNF-α is the main regulatory cytokine in both RA and periodontitis. TNF-α inhibitors (anti-TNF-α) reduce the number of inflammatory cells, osteoclast formation and bone loss. In addition, many immunological processes have been identified that are similar to both diseases. Autoreactive T cells, natural killer cells, heat shock proteins, autoantibodies and genetic factors are reported to play an important role in the inflammatory pathway of RA and periodontitis.

Recently, TNF-α blocking agents (anti-TNF-α) have been developed and used for the treatment of RA. Animal and human studies have suggested that anti-TNF-α treatment may reduce the severity of periodontitis.

The aim of this study was to investigate the effect of nonsurgical periodontal treatment combined with anti-TNF-α on alveolar bone loss and oxidative stress in individuals with RA and periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Having a confirmed diagnosis of Rheumatoid Arthritis (RA),
* Having a diagnosis of Stage III-IV periodontitis,
* Having at least 20 teeth,

Exclusion Criteria:

* Having used antibiotics for the 3 months before the study,
* Being pregnant and lactating,
* Having received periodontal treatment in the last 6 months,
* Being diabetic.
* Smoking.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Periodontal pocket depth | baseline, 3rd month after non-surgical periodontal therapy, 6th month after non-surgical periodontal therapy
  The distance between the pocket base and the gingival margin is measured
clinical attachment loss | baseline, 3rd month after non-surgical periodontal therapy, 6th month after non-surgical periodontal therapy
  The distance between the pocket base and the cementoenamel junction is measured

SECONDARY OUTCOMES:
serum and GCF receptor activator nuclear kappa B ligand (RANKL) level | baseline, after non-surgical periodontal therapy at 3 months, after non-surgical periodontal therapy at 6 months,
  RANKL levels in serum and GCF will be measured with biochemical kits.
serum and GCF osteoprotegrin (OPG) level | baseline, after non-surgical periodontal therapy at 3 months, after non-surgical periodontal therapy at 6 months,
  OPG levels in serum and GCF will be measured with biochemical kits.
serum and GCF matrix metalloproteinase 8 (MMP8) level | baseline, after non-surgical periodontal therapy at 3 months, after non-surgical periodontal therapy at 6 months,
  MMP-8 levels in serum and GCF will be measured with biochemical kits.
serum total antioxidant status (TAS) level | baseline, after non-surgical periodontal therapy at 3 months, after non-surgical periodontal therapy at 6 months,
  TAS levels in serum will be measured with biochemical kits.
serum total oxidant status (TAS) level | baseline, after non-surgical periodontal therapy at 3 months, after non-surgical periodontal therapy at 6 months,
  TOS levels in serum will be measured with biochemical kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Dentistry, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The requested data can be shared in a way that protects patient personal information.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year as of 02.02.2025

REFERENCES:
- [Background] de Pablo P, Dietrich T, McAlindon TE. Association of periodontal disease and tooth loss with rheumatoid arthritis in the US population. J Rheumatol. 2008 Jan;35(1):70-6. Epub 2007 Nov 15. PMID 18050377